CLINICAL TRIAL: NCT03284450
Title: Exercise Induced Muscle Damage Post Dance and Sprint Specific Exercise in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Glyn Howatson, Reader - Human and Applied Physiology, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NUMB1
Record Dates: First submitted 2016-09-28; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Exercise Induced Muscle Damage
Keywords: Dance; Sprint; Females; Recovery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dance performance fitness test (DPFT) (Experimental)
  Interventions: Other: DPFT
- Sport specific repeated sprints (SSRS) (Active Comparator)
  Interventions: Other: SSRS

INTERVENTIONS:
Other: DPFT — The DPFT described previously (Redding et al., 2009) involves the repetition of a 'dance phrase' representative of contemporary dance, with each phrase separated by a 2 minute rest period. For the present study the originally described test was extended; the adapted protocol involved 10 x 1 minute movement phrases, each separated by 2 minutes rest.
  Arms: Dance performance fitness test (DPFT)
Other: SSRS — The SSRS (Howatson & Milak, 2009) involved 15 x 30 m sprints with a rapid 10 m deceleration phase, with each sprint departing every 65 seconds.
  Arms: Sport specific repeated sprints (SSRS)

SUMMARY:
There is a paucity of studies investigating exercise-induced muscle damage (EIMD) in females and only one in response to dance-type exercise. This study aimed to firstly elucidate the physiological profile of EIMD following a dance-specific protocol, and second to compare the magnitude of damage to that experienced following a sport-specific protocol in physically active females.

DETAILED DESCRIPTION:
Twenty nine female recreational dancers from a University dance team volunteered to take part in the study. A 3-day food diary and activity log completed prior to testing determined that there were no differences in physical activity levels or energy and macronutrient intakes between participants. Subjects were asked to replicate their reported diets as closely as possible throughout the testing period. A menstrual cycle questionnaire was also completed in order to determine menstrual cycle phase; all testing took place during the early/mid luteal phase.

Participants were randomly assigned to two exercise groups designed to induce EIMD; either a dance-specific protocol (DPFT) or a sport-specific repeated sprint protocol (SSRS). Participants completed the DPFT (n=15) or SSRS (n=14) and a battery of commonly used muscle damage indices were measured pre, immediately post and 24-, 48-, and 72 h post muscle damage. These were; delayed onset muscle soreness (DOMS), limb girth, countermovement jump height (CMJ), reactive strength index (RSI), maximal voluntary isometric contraction (MVC) sprint performance, and total creatine kinase (CK) activity. Participants were tested at the same time on subsequent days (± 1 h) to account for diurnal variation. Participants were asked to avoid strenuous exercise, alcohol, caffeine, nutritional supplements and any anti-inflammatory drugs or alternative treatments for the duration of the study.

Statistical software (IBM SPSS v21, IBM, USA) was used for inferential analysis and significance was accepted at the P < .05 a priori. Mauchley's test assessed the sphericity of the data and where appropriate, violations were corrected using the Greenhouse-Geisser. To explore our first objective, a one-way analysis of variance (ANOVA) with repeated measures (group, 1; time, 5) was performed on all variables in order to analyse the muscle damage response to the DPFT. For the second aim a two-way ANOVA with repeated measures (group, 2; time, 5) was used for all variables to allow for comparison of the muscle damage response between the DPFT and the SSRS. Where appropriate LSD post-hoc analysis was performed.

ELIGIBILITY:
Inclusion Criteria:

* physically active
* at least 3 years experience in dance training

Exclusion Criteria:

* presence of any medical or physical conditions, either chronic or sustained in the last 3 months which would make participation difficult or harmful to the participant
* eg. history of cardiovascular disease and musculoskeletal disorders

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in maximum voluntary contraction (MVC) | Change from pre exercise MVC at 24 h post exercise
  Isometric MVC of the participants' dominant knee extensors was assessed using a strain gauge.

SECONDARY OUTCOMES:
Limb girths | pre, immediately post (0) and 24-, 48-, and 72 h post exercise
  Lower limb girths at the calf and mid-thigh of the right leg were recorded as measures of muscle swelling. Both locations were marked with permanent marker to ensure consistency on consecutive days.
Countermovement jump | pre, immediately post (0) and 24-, 48-, and 72 h post exercise
  Countermovement jump height was recorded using a light timing system.
Reactive strength index | pre, immediately post (0) and 24-, 48-, and 72 h post exercise
  Participants performed a drop jump from a 30cm height to determine reactive strength index
Muscle soreness | pre, immediately post (0) and 24-, 48-, and 72 h post exercise
  Subjective muscle soreness was measured using a 200 mm visual analogue scale from 'no soreness' to 'unbearably sore.' Participants were required to indicate on the line the level of perceived active lower limb soreness felt during a 90 degree squat.
30 m sprint time | pre, immediately post (0) and 24-, 48-, and 72 h post exercise
  Participants completed a single maximal effort 30 m sprint where sprint time was recorded. The sprint was initiated from a line 30 cm behind the start line in order to prevent false triggering of the timing gates.
Creatine Kinase | pre, immediately post (0) and 24-, 48-, and 72 h post exercise
  Blood samples were collected via venepuncture from the antecubital fossa area in to a 10 ml EDTA vacutainer. The samples were centrifuged at 3000 RCF for 15 minutes at 4 C. Plasma was extracted, and stored immediately at -80 C for later analysis. Plasma CK concentrations were determined spectrophotometrically.

CONTACTS AND LOCATIONS:
Overall Officials: Emma J Stevenson, PhD, Principal Investigator — Northumbria University